CLINICAL TRIAL: NCT07239310
Title: A Prospective, Multicenter, Randomized, Double-Blind, Parallel-Group, Confirmatory Clinical Trial to Verify the Efficacy and Safety of the Cognitive Improvement Effect on Executive Function in Medication-Treated Patients With Mild Cognitive Impairment and Prodromal Alzheimer's Disease Using the Neuclare Physical Device for Medical Use
Brief Title: Neuclare Device for Temporary Improvement of Executive Function in Patients With Mild Cognitive Impairment and Prodromal Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deepsonbio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-Altheon; 1861 (Other: Ministry of Food and Drug Safety (MFDS))
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease(AD)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Neuclare Device (Experimental): Participants receive standard medication plus Neuclare device therapy three times per week for 4 weeks.
  Interventions: Device: Participants receive Neuclare Device while continuing their cognitive medication
- Sham Device (Placebo Comparator): Participants receive standard medication plus sham Neuclare device therapy.
  Interventions: Device: Participants receive Sham Neuclare Device while continuing their cognitive medication

INTERVENTIONS:
Device: Participants receive Neuclare Device while continuing their cognitive medication — Participants in this arm receive the Neuclare physical device applied to the cerebral cortex, receiving low-intensity ultrasound stimulation less than 30 minutes per session, three times per week for 4 weeks.
  This intervention is intended to temporarily improve executive function in patients with mild cognitive impairment and prodromal Alzheimer's disease.
  Arms: Neuclare Device
Device: Participants receive Sham Neuclare Device while continuing their cognitive medication — Participants in this arm receive a sham version of the Neuclare device, which mimics the appearance and procedure of the active device but does not deliver therapeutic ultrasound.
  The sham device is applied less than 30 minutes per session, three times per week for 4 weeks, while participants continue their cognitive medication.
  This arm serves as a control for comparison with the active intervention.
  Arms: Sham Device

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel-group, prospective confirmatory clinical trial designed to evaluate whether the Neuclare medical device can temporarily improve executive function (planning and problem-solving abilities) in adults with mild cognitive impairment or very early Alzheimer's disease.

Participants will continue their current medication and be randomly assigned to receive either the Neuclare device (treatment group) or a sham device (control group). The device will be applied to the brain three times per week for four weeks. Both participants and study staff are blinded to the group assignment. Safety and adverse events will be closely monitored throughout the study.

During the trial, assessments will include attention, cognitive function, daily living activities, brain imaging (Amyloid PET-CT), blood biomarkers, and quality of life (EQ-5D-5L).

The goal of this study is to determine whether the Neuclare device, in combination with standard medication, can safely provide temporary improvements in executive function.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 55 to 90 years.
2. Diagnosed with probable Alzheimer's disease according to NINCDS-ADRDA criteria and DSM-IV criteria for dementia,
3. or mild cognitive impairment/very mild Alzheimer's disease with CDR 0.5-1 and MMSE-II ≥18.
4. On stable cognitive therapy medications for at least 1 month.
5. Voluntary participation with signed informed consent.

Exclusion Criteria:

1. Patients with structural brain lesions detected on brain MRI (e.g., cerebral edema, intracerebral hemorrhage, cerebral infarction, cerebrovascular malformation, brain tumor, etc.).
2. Patients with uncontrolled metabolic disorders such as thyroid dysfunction, hypoglycemia, or hepatic/renal impairment, or those on long-term medications that may cause cognitive impairment (e.g., anticholinergic drugs).
3. Patients with a history of epileptic seizures, depression, or psychiatric disorders; patients experiencing visual hallucinations or fluctuating cognitive decline.
4. Patients with psychiatric disorders outside of the inclusion criteria.
5. Patients with a history of severe diseases such as cancer or tuberculosis.
6. Patients with a history of or currently taking psychoactive drugs or medications affecting the central or peripheral nervous system.
7. Patients with contact dermatitis or other skin hypersensitivity conditions.
8. Patients with fever ≥ 40°C as measured by tympanic temperature.
9. Patients who have experienced bleeding within the past 3 months due to procedures or surgeries that may affect vital signs.
10. Patients unable to undergo MRI.
11. Pregnant patients.
12. Patients with clinical brain calcification observed on computed tomography (CT) scans.
13. Patients with known allergies to contrast agents such as Definity or Gadovist.
14. Any other condition deemed by the investigator to make participation in the clinical trial inappropriate.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Trail Making Test-A Completion Time from Baseline to Week 5 | 5 weeks
  The primary efficacy outcome is the change in Trail Making Test-A (TMT-A) completion time from baseline to Week 5 after application of the investigational device. Descriptive statistics will be presented for each treatment arm. Between-group comparisons of the change from baseline will be analyzed using ANCOVA with baseline scores as a covariate.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ewha Womans University Mokdong Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No